CLINICAL TRIAL: NCT05994612
Title: Suicide Prevention for Substance Using Youth Experiencing Homelessness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023B0145
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Therapy for Suicide Prevention + Services as Usual (Experimental): 10 sessions of Cognitive Therapy for Suicide Prevention (CTSP) provided over 6 months, with 9 optional booster sessions + services as usual (SAU) received by the community.
  Interventions: Behavioral: Cognitive Therapy for Suicide Prevention; Behavioral: Services as Usual
- Services as Usual (Active Comparator): Services as Usual involves utilizing Strengths-Based Outreach and Advocacy to link youth to community services for a period of 6 months.
  Interventions: Behavioral: Services as Usual

INTERVENTIONS:
Behavioral: Cognitive Therapy for Suicide Prevention — 10 sessions of cognitive therapy for suicide prevention plus 9 optional booster sessions
  Other Names: CTSP
  Arms: Cognitive Therapy for Suicide Prevention + Services as Usual
Behavioral: Services as Usual — Participants will receive services that they would normally receive in the community.
  Other Names: SAU

SUMMARY:
Suicide is the leading cause of death among YEH and most youth do not access services that may be available to them. Therefore, this study seeks to address this gap in the research literature with the goal to identify an effective intervention that can be readily adopted by communities that serve these youth. We will test the effects of outreach-worker delivered Cognitive Therapy for Suicide Prevention (CTSP)+Services as Usual (SAU) versus SAU alone on suicidal ideation (primary outcome), substance use and depressive symptoms (secondary outcomes) at 3, 6, 9 and 12- months.

DETAILED DESCRIPTION:
While research on substance using youth experiencing homelessness (YEH) is increasing, there is a dearth of information regarding effective prevention interventions for these youth. This is of significant concern because studies indicate that 66% to 89% of YEH have a mental health disorder and 68% report at least one suicide attempt . In fact, suicide is the leading cause of death among YEH. Among those who have attempted suicide, an average of 6.2 attempts is reported, and lifetime suicidal ideation rates range from 14% to 66.5% with no clear evidence of effective interventions for YEH. This study uses general cognitive theory, complemented with concepts from two suicide specific theoretical models, to guide our intervention and conceptual change model. The study goal is to test strategies to extend delivery and uptake of a cognitive therapy intervention for YEH. Prior studies focus on service-connected youth, but research suggests that most street living YEH do not access services meant to assist them. Prior sampling limitations are overcome through engaging service-disconnected youth in addition to service-connected youth through a local drop-in center. As such, three hundred substance using YEH with recent suicidal ideation or a recent suicide attempt will be randomly assigned to Cognitive Therapy for Suicide Prevention (CTSP) + Services as Usual (SAU) (N=150) or to SAU alone (N=150). CTSP has previously shown efficacy for YEH through a RCT pilot feasibility study. SAU includes outreach, advocacy and service linkage which are typical services offered by agencies serving those experiencing homelessness. Follow-up assessments will be conducted at 3, 6, 9 and 12-months post-baseline. It is hypothesized that youth receiving CTSP+SAU will show greater reductions in suicidal ideation (primary outcome), substance use and depressive symptoms (secondary outcomes) over time compared to SAU alone, as well as improved risk and protective factors. Theoretically-derived mediators will be tested to shed light on mechanisms associated with change, and the moderating effects of sex, race, sexual orientation and baseline service connection will be examined. In order to ease future dissemination of the intervention to agencies serving YEH, the investigators will rigorously assess acceptability, feasibility, fidelity and cost associated with the delivery of our intervention approach using a mixed-methods approach. Ultimately, the goal of this research is to provide support for the use of a suicide prevention intervention for substance using YEH that reduces premature mortality, hospitalization, and loss of human capital and which can be easily adopted by agencies serving YEH.

ELIGIBILITY:
Inclusion Criteria:

* 15-24 years
* SSI-W score > 4 or at least one suicide attempt in prior 12 months
* Meets criteria for homelessness
* At least four uses of alcohol/drugs in prior 30 days

Exclusion Criteria:

* Youth requires psychiatric hospitalization

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation: Scale for Suicidal Ideation-Worst Point (SSI-W) | baseline, 3, 6, 9 and 12 months
  Change in suicidal ideation is measured using the Scale for Suicidal Ideation-Worst Point (SSI-W). Each item consists of three options, which are rated on a 3-point scale from 0 to 2, and each item is graded according to the intensity of the suicidality. Total scores are calculated by summing the 19 ratings, and these total scores can range from 0 to 38 with higher scores indicating worse severity.

SECONDARY OUTCOMES:
Depressive Symptoms: Beck Depression Inventory II | baseline, 3, 6, 9 and 12 months
  The Beck Depression Inventory II is a 21-item inventory that assesses the severity of depressive symptomatology. Each item is rated on a 0-3 scale with summary scores ranging between 0 and 63 and higher scores indicating higher depressive symptomatology.
Substance use: Form 90 | baseline, 3, 6, 9 and 12 months
  Frequency of substance use is measured using the Form-90, a semi-structured questionnaire that uses the timeline follow-back method. Form yields percentage of days in the prior 90 days using alcohol and drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Slesnick, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share results from surveys after de-identification through the Inter-University Consortium for Political and Social Research (ICPSR), an NIH funded data repository, within one year of completion of data collection (see https://www.icpsr.umich.edu/icpsrweb/). Submitted data will conform with relevant data and terminology standards.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: one year after project close-out.
Access Criteria: Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) for secondary study/data analysis purposes and with study PI approval.

REFERENCES:
- [Derived] Slesnick N, Brakenhoff B, Chavez LJ, Cuthbertson CL, Famelia R, Feng X, Ford J, Holowacz E, Jaderlund S, Kelleher K, Luthy E, Mallory AM, Pizzulo A, Slesnick TD, Yilmazer T. Suicide prevention for substance using youth experiencing homelessness: study protocol for a randomized controlled trial. Trials. 2024 Mar 9;25(1):174. doi: 10.1186/s13063-024-07997-y. PMID 38461275